CLINICAL TRIAL: NCT06023121
Title: Use of a Liquid Biopsy Signature as Blood Biomarker for Early Detection and Monitoring Early-onset Gastric Cancer
Brief Title: Use of a Liquid Biopsy Signature to Detect Early-onset Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Lin Chen, Director of department of General Surgery, Chinese PLA General Hospital
Other Study IDs: EOGC-biomarker
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Gastric cancer cases from two medical centers in China
  Interventions: Diagnostic Test: Measurement of levels of an exosome-based liquid biopsy signature
- Controls: Controls from two medical centers in China
  Interventions: Diagnostic Test: Measurement of levels of an exosome-based liquid biopsy signature

INTERVENTIONS:
Diagnostic Test: Measurement of levels of an exosome-based liquid biopsy signature — Each participant was enrolled to assess the levels of an exosome-based liquid biopsy signature

SUMMARY:
Early-onset gastric cancer (EOGC) is a lethal malignancy with a poor prognosis. It differs from late-onset gastric cancer (LOGC) in clinical and molecular characteristics. The current strategies for EOGC detection have certain limitations in diagnostic performance due to the rising trend in EOGC. Hence, identifying novel EOGC bioindicators is crucial.

DETAILED DESCRIPTION:
Due to widespread gastric cancer (GC) detection efforts and timely interventions (removal of precancerous lesions and early-stage GC), the GC-associated mortality rate has declined worldwide. However, epidemiological studies show rising GC incidences among young adults (< 50 years old) without familial or hereditary origin. This illness, known as early-onset GC (EOGC), comprises 20-30% of new GC diagnoses, mainly among individuals aged 30-40 years; the median overall survival time is 11.7 months. Although the underlying cause behind this trend is poorly understood, there is a general understanding that EOGC epidemiologically, biologically, and pathologically differs from late-onset GC (LOGC, ≥ 50 years). Therefore, EOGC patients require clinical assessment and intervention distinct from those applied in LOGC.

Of note, several population-based epidemiological studies have suggested that EOGC patients exhibit significantly different behaviors from LOGC patients. EOGC patients are more likely to have earlier lymph node and distal metastasis than LOGC patients during disease progression. These tough challenges raise clinical concerns: EOGC is more aggressive than LOGC; thus, a delayed diagnosis can severely affect patient survival outcomes. Moreover, the current approaches to GC detection, such as CEA, HP serology, and pepsinogen (PG), are insufficient for detecting early-stage GC and have yet to be investigated in young individuals with EOGC. Accordingly, these limitations strongly underscore the necessity to establish potent alternative indicators that facilitate the timely detection of EOGC.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* 50 years old ≥ Age ≥ 18 years old
* Histologically confirmed gastric adenocarcinoma

Exclusion Criteria:

* Other previous malignancy within 5 year
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study
* Pregnancy or lactation period
* Legal incapacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample Shanxi - Hospital and community sample Beijing -Hospital
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Detection of levels of an exosome-based liquid biopsy signature | Through study completion, an average of 3 year
  A three exo-LR (NALT1, PTENP1, and HOTTIP) liquid biopsy signature was developed for EOGC detection.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital Ethics Committee, Beijing, Beijing Municipality, China